CLINICAL TRIAL: NCT00486031
Title: A Multicenter, Open-label Trials to Evaluate the Long-term Safety and Tolerability of a New Balsalazide Disodium Tablet Formulation in Patients With Ulcerative Colitis
Brief Title: Open-Label, Long-term Balsalziade Disodium Tablet Ulcerative Colitis Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BZUC3005
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: IBD; UC; Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — balsalazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- balsalazide disodium tablets,3.3 g BID, (Other)
  Interventions: Drug: Balsalazide Disodium

INTERVENTIONS:
Drug: Balsalazide Disodium

SUMMARY:
The objective of the study is to evaluate the long-term safety and tolerability of treatment with balsalazide disodium tablets in subjects who are in remission from ulcerative colitis or who have mildly to moderately active UC.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the long-term safety and tolerability of treatment with balsalazide disodium tablets in subjects who are in remission from ulcerative colitis or who have mildly to moderately active UC.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a documented history of UC and is either in remission or currently presents with mildly to moderately active UC symptoms as determined by the investigator upon subject interview of UC symptoms, (e.g., urgency, bowel frequency, and rectal bleeding). Additionally, the diagnosis of UC must be confirmed by past flexible sigmoidoscopy/colonoscopy which may include colonic mucosal pathological findings on biopsy consistent with UC.
* Subject is capable and willing to comply with all study procedures.

Exclusion Criteria:

* Subject has a history of allergy or intolerance to aspirin, mesalamine or other salicylates.
* Subject has participated in an investigational drug or device study, other than a previous balsalazide disodium tablet trial (i.e., BZUC3002 or BZUC3003), within 30 days of entering the current study.
* Subject discontinued from a previous balsalazide disodium tablet study due to study drug-related AE(s), including UC flare or associated symptoms that were perceived by the subject/investigator as being caused by study drug.
* Subject has had any prior bowel surgery, except appendectomy and cholecystectomy.
* Subject has unstable cardiovascular, coagulopathy, or pulmonary disease.
* Regular use of nonsteroidal anti-inflammatory drugs (NSAIDS) except cardioprotective ASA (i.e., less than or equal to 162 mg ASA per day).
* Subject has a history of human immunodeficiency virus (HIV) or hepatitis (B and C). Subjects with a history of hepatitis B and C will be eligible provided the screening LFTs are within normal limits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (95):
  - Birmingham Gastroenterology Associates, PC, Birmingham, Alabama
  - Premeire Pharmaceutical Research, Tempe, Arizona
  - Medical Services of NWA, Fayetteville, Arkansas
  - AGMG Clinical Research Institute, Anaheim, California
  - Discovery Clinical Research, Inc., Encinitas, California
  - Digestive and Liver Disease Specialists, Garden Grove, California
  - West Gastroenterology Medical Group, Los Angeles, California
  - Community Clinical Trials, Orange, California
  - Sharp Rees-Stealy Medical, San Diego, California
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Arapahoe Gastrroenterology, PC, Littleton, Colorado
  - South Denver Gastroenterology, Lone Tree, Colorado
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Clinical Trials Management of Boca Raton, Boca Raton, Florida
  - Research Consultants Group, Hialeah, Florida
  - Horizon Institute for Clinical Research, Hollywood, Florida
  - Mark Lamet, M.D., Hollywood, Florida
  - Southern Clinical Research Consultants, Hollywood, Florida
  - A+ Research, Miami, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Venture Research Institute, LLC, North Miami Beach, Florida
  - West Wind'r Research & Development, Tampa, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Dekalb Gastroenterology Associates, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Digestive Research Associates, Newnan, Georgia
  - University Digestive Health Center, Oak Forest, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Iowa Digestive Disease Center, PC, Clive, Iowa
  - Cotton-O'Neil Digestive Health Center, Topeka, Kansas
  - Digestive Health Center of Louisiana, Baton Rouge, Louisiana
  - Clinical Trials Management, Metairie, Louisiana
  - Digestive Disorders Associates, Annapolis, Maryland
  - Alan Rosen, M.D., Baltimore, Maryland
  - Digestive Disease Association, Baltimore, Maryland
  - Metro Gastroenterology Group, Chevy Chase, Maryland
  - Washington County Hospital, Hagerstown, Maryland
  - Philip J. Bean Medical Center, Hollywood, Maryland
  - Charm City Research, Lutherville, Maryland
  - Coastal Research Associates, Inc., Braintree, Massachusetts
  - Clinical Research Institute of Michigan LLC, Chesterfield, Michigan
  - Gastroenterology Associates of West Michigan, Grand Rapids, Michigan
  - Gastrointestinal Associates, Jackson, Mississippi
  - Center for Digestive and Liver Diseases, Mexico, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Central Jersey Medical Research, Elizabeth, New Jersey
  - Shore Health Group, Ocean City, New Jersey
  - The GI Group of South Jersey, Vineland, New Jersey
  - Long Island Clinical Research, Great Neck, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York
  - Simon Lichtiger, MD, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Charlotte Gastroenterology & Hepatology, Charlotte, North Carolina
  - Northwest Piedmont Clinical Research, Elkin, North Carolina
  - LeBauer Research Associates, PA, Greensboro, North Carolina
  - Carolina Digestive Diseases, PA, Greenville, North Carolina
  - East Carolina Gastroenterology, PA, Jacksonville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Gastroenterology Specialists, Inc., Canton, Ohio
  - Consultants for Clinical Research, Inc., Cincinnati, Ohio
  - Digestive Health Newtork, Cincinnati, Ohio
  - Gastrointestinal & Liver Disease Consultants, Dayton, Ohio
  - Avamar Center for Endoscopy, Warren, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - George Koval, M.D., Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Guthrie Clinic, Ltd, Sayre, Pennsylvania
  - Charleston Gastroenterology Center, Charleston, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Memphis Gastroenterology Group, Memphis, Tennessee
  - Gastrointestinal Institute, PLLC, Nashville, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Austin Gastroenterology, Austin, Texas
  - NationsMed Clinical Research, Houston, Texas
  - Houston Digestive Diseases Clinic, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - Baylor University Medical Center, Irving, Texas
  - North Texas Gastroenterology, Lewisville, Texas
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - McGuire VAMC, Richmond, Virginia
  - Seattle Gastroenterology Associates, Seattle, Washington
  - Tacoma Digestive Disease Research, Tacoma, Washington
  - Discovery Research International, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Balsalazide Disodium Tabs,3.3 g BID: Balsalazide Disodium tablets,3.3 g BID
Period: Overall Study
Arm/Group | Balsalazide Disodium Tabs,3.3 g BID
Started | 443
Completed | 440
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Balsalazide Disodium Tabs,3.3 g BID,: balsalazide disodium tablets,3.3 g BID,
Arm/Group | Balsalazide Disodium Tabs,3.3 g BID,
Number analyzed (Participants) | 440
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 412
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 224

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent AEs
Description: Incidence of treatment emergent adverse events
Time Frame: 24 Months
Measure: Number; unit: participants
Groups:
- Balsalazide Disodium: balsalazide disodium tablets,3.3 g BID,
Arm/Group | Balsalazide Disodium
Number analyzed (Participants) | 440
participants | 273

2. Secondary Outcome: Time to Onset of AEs
Description: Time to onset of adverse events
Time Frame: 24 Months
Population: Data were not collected to perform this analysis
Arm/Group | Balsalazide Disodium Tabs,3.3 g BID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Balsalazide Disodium
Serious Adverse Events (participants affected / at risk) | 21/440
Other Adverse Events (participants affected / at risk) | 273/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Balsalazide Disodium (N=440)
Colitis ulcerative (Gastrointestinal disorders) | 5
ANAEMIA (Blood and lymphatic system disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CHEST PAIN (Cardiac disorders) | 1
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
APPENDICITIS (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
CLOSTRIDIAL INFECTION (Infections and infestations) | 1
CLOSTRIDIUM COLITIS (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
PANCREATIC ENZYMES INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Balsalazide Disodium (N=440)
Worsening UC (Gastrointestinal disorders) | 48
Diarrhea (Gastrointestinal disorders) | 27
Abdominal pain (Gastrointestinal disorders) | 26
Rectal haemorrhage (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 13
Abdominal tenderness (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 8
Hematochezia (Gastrointestinal disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 7
Urinary tract infection (Infections and infestations) | 21
Nasopharyngitis (Infections and infestations) | 19
Upper respiratory tract infection (Infections and infestations) | 19
Sinusitis (Infections and infestations) | 15
Influenza (Infections and infestations) | 13
Bronchitis (Infections and infestations) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 8
Headache (Nervous system disorders) | 24
Dizziness (Nervous system disorders) | 8
Insomnia (Product Issues) | 8
Depression (Psychiatric disorders) | 7
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Rash (Respiratory, thoracic and mediastinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes